CLINICAL TRIAL: NCT01983189
Title: Repetetive Transcranial Magnetic Stimulation for Evaluation and Treatment of Repetetive Behavior in Subjects With Autism Spectrum Disorders.
Brief Title: Transcranial Magnetic Stimulation for Evaluation and Treatment of Repetetive Behaviors in Autism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal investigator (Dr. Sporn) left the sponsoring institution.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 5594
Record Dates: First submitted 2012-03-14; First posted 2013-11-13 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-01

CONDITIONS: Autism; Asperger Disorder; Other Developmental Pervasive Disorder
Keywords: TMS; transcranial magnetic stimulation; rTMS; recurrent transcranial magnetic stimulation; fMRI; functional magnetic resonance imaging.
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low frequency rTMS (Experimental): low frequency, repetitive transcranial magnetic stimulation (rTMS) for 20 minutes daily, 5 times a week for 3 weeks
  Interventions: Procedure: transcranial magnetic stimulation

INTERVENTIONS:
Procedure: transcranial magnetic stimulation — 1 hz transcranial magnetic stimulation

SUMMARY:
This study is a trial of low frequency Repetitive Transcranial magnetic stimulation( rTMS) for subjects with autism spectrum disorders, specially targeting repetitive behaviors.

DETAILED DESCRIPTION:
This project is a 3-week double blind cross-over trial for adolescents and adults who meet criteria for autism and have clinically prominent repetitive behaviors. The investigator will apply low frequency rTMS for 20 minutes 5 times a week for 3 weeks targeting the area of brain which was involved in repetitive behaviors. The investigator will obtain clinical measures of repetitive behaviors as well as social functioning pre and post treatment. As a control and a cross-over condition , we will stimulate other area of brain which has nothing to do with repetitive behaviors but may improve social functioning in autism spectrum disorders. In addition to r TMS we will perform a pre and post treatment perfusion functional MRI and obtain TMS measure of excitability of brain.

ELIGIBILITY:
Inclusion Criteria:

1. English Speaking
2. Capacity to give consent and sign HIPAA Authorization
3. Patients currently taking psychotropic medications must be at the same stable dose and likely to be able to continue at the same dose throughout the study
4. ASD diagnosis according to the DSM-IV TR Symptom and Criterion checklist for ASD
5. Significant level of repetitive behaviors to distinguish from movement disorders to be in at least 3 out of 6 sub-scales (stereotyped behavior, self-injurious behavior, compulsive behavior, ritualistic behavior, sameness behavior, restricted behavior) -

Exclusion Criteria:

1. Women of child-bearing potential not using birth control, pregnant or breast feeding
2. H/o Bipolar Disorder (lifetime), any Psychotic Disorder (lifetime) history of Major Depressive Disorder or of substance abuse or dependence within the past year
3. Significant sub-average intellectual function (IQ<70)
4. Intracranial implants
5. Increased risk of seizure for any reason, including prior diagnosis of epilepsy, seizure disorder, febrile seizure, increased intracranial pressure or history of significant head trauma with loss of consciousness for > 5 minutes.
6. Current significant laboratory abnormality
7. Neurological disorder including but not limited to space occupying brain lesion, any history of seizures, history of cerebrovascular accident, fainting, cerebral aneurysm, dementia, Huntington chorea, Multiple Sclerosis -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
clinical improvement based on repetitive behavior scale. | baseline-week3

SECONDARY OUTCOMES:
clinical improvement based on the social responsiveness scale. | before-week3

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Sporn, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, United States